CLINICAL TRIAL: NCT04718675
Title: Phase 1, First-in-human, Open-label Dose Escalation and Cohort Expansion Study of KB-0742 in Patients With Relapsed or Refractory Solid Tumors or Non-Hodgkin Lymphoma
Brief Title: A Study of KB-0742 in Participants With Relapsed or Refractory Solid Tumors Including Platinum Resistant High Grade Serous Ovarian Cancer (HGSOC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to lack of safety and futility
Sponsor: Kronos Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB-0742-1001; 2023-503739-16-00 (Other: EU CT Number)
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Relapsed Solid Tumors; Refractory Solid Tumors; Non-Hodgkin Lymphoma; HGSOC; Platinum Resistant High Grade Serous Ovarian Cancer
Keywords: KB-0742; Relapsed Solid Tumors; Refractory Solid Tumors; Non-Hodgkin Lymphoma; CDK9 Inhibitor; Platinum Resistant High Grade Serous Ovarian Cancer; HGSOC; BRCA1 mutation; BRCA2 mutation; HRD positive; MYC amplification/overexpression
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Sequential cohorts of participants will receive escalating doses of KB-0742.
  Interventions: Drug: KB-0742
- Part 2: Cohort Expansion (Experimental): Following identification of the contingent recommended Phase 2 dose (RP2D) in Part 1, the following expansion cohorts will be enrolled:
  Cohort A: Participants with R/R non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC), and high grade serous ovarian cancer.
  Cohort B: Participants with R/R small cell lung cancer (SCLC), NUT midline carcinomas (NMC), adenoid cystic carcinoma (ACC), chordoma and soft tissue sarcomas associated with transcription factor fusion.
  Interventions: Drug: KB-0742

INTERVENTIONS:
Drug: KB-0742 — Oral capsules

SUMMARY:
Part 1: Dose Escalation. The primary objective of Part 1 of this study is to evaluate the safety and tolerability of KB-0742 in participants with relapsed or refractory (R/R) solid tumors or non-Hodgkin lymphoma (NHL).

Part 2: Cohort Expansion. The primary objective of Part 2 of this study is to further evaluate the safety and tolerability of KB-0742 in defined participant cohorts including Platinum Resistant High Grade Serous Ovarian Cancer (HGSOC).

DETAILED DESCRIPTION:
Part 2 cohort expansion is now enrolling Platinum Resistant High Grade Serous Ovarian Cancer (HGSOC) patients who may have one or more of these genetic alterations, BRCA 1 mutation, BRCA 2 mutation, MYC amplification/ overexpression, Homologous Recombination Deficient (HRD) positive.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 18 years old (Parts 1 and 2A); males or females ≥ 12 years old and with a body weight ≥ 40 kg are eligible to enroll with tumor types including soft-tissue sarcomas, Ewing's sarcoma, alveolar rhabdomyosarcoma, NUT midline carcinoma (NMC), or chordoma (Part 2B)
* Willing and able to provide consent (and assent for participants between the ages of 12 to <18)
* Part 1: Participants who meet at least 1 of the following criteria:

  1. Any R/R solid tumor with, in the opinion of the investigator at the time of screening has at least 1 readily accessible biopsy site(s) and who consents to 1 baseline and 1 on-treatment biopsy. If the feasibility of obtaining biopsies changes after the participant has been consented due to changes in clinical or surgical considerations and the participant otherwise meets all eligibility criteria, they may still enroll/or continue on study.
  2. Tumor type of interest (see list below) with measurable disease per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST) 1.1 or Positron Emission Tomography (PET) Response Criteria in Solid Tumors (PERCIST) 1.0 for solid tumors or by Lugano Classification or Modified Weighted Assessment Tool (mSWAT) for NHL AND at least 1 measurable scan per one of the above criteria prior to the most recent scan to document the rate of tumor growth before the initiation of study treatment. Tumor types of interest (R/R without other available therapeutic options) are:

     1. SCLC
     2. Epithelial ovarian cancer, TNBC, or NSCLC
     3. Other epithelial solid tumor with evidence of MYC copy number gain based on local testing
     4. Diffuse large B-cell lymphoma with documented MYC translocation or Burkitt's lymphoma (as determined by local testing)
     5. Sarcoma of histologic subtypes known to be associated with transcription factor fusion, specifically: i. Myxoid/round cell sarcoma ii. Clear cell sarcoma iii. Desmoplastic small round cell tumor iv. Low grade fibromyxoid sarcoma v. Extraskeletal myxoid chondrosarcoma vi. Ewing sarcoma vii. Alveolar rhabdomyosarcoma
     6. Chordoma, NUT midline carcinoma, or adenoid cystic carcinoma
* Part 2, Cohort A: Participants with histologically or cytologically confirmed solid tumors who have failed, are intolerant to, or are considered ineligible for standard-of-care anti-cancer treatments. Note: Part 2, Cohort A, will include participants with relapsed or refractory solid tumors including NSCLC, TNBC and ovarian cancer.
* Part 2, Cohort B: Participants with histologically or cytologically confirmed tumor type of interest without access to or intolerant of other approved therapies, including SCLC.
* For both Parts 1 and 2:
* Access to a tumor sample for central laboratory testing
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1
* Evaluable or measurable disease, per RECIST 1.1 or PERCIST 1.0 for solid tumors or the Lugano Classification or mSWAT for NHL
* Adequate bone marrow and organ function
* Recovery from treatment-related toxicities from prior therapies to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade ≤ 1 or to baseline level
* Must agree to use highly effective birth control during the trial and for at least 3 months after the last dose of study drug; female participants cannot be pregnant or breastfeeding

Exclusion Criteria:

* Any other anti-cancer therapies including chemotherapy, immunotherapy, or hormonal therapy within 4 weeks or 5 half-lives (whichever is shorter)
* History of surgery (except for diagnostic purposes) or non-palliative radiotherapy within 4 weeks
* History of allogeneic transplantation within 6 months
* Active central nervous system (CNS) involvement by the underlying malignancy; previously treated CNS metastatic disease is permitted with magnetic resonance imaging (MRI) documentation of stable disease for at least 3 months prior to study start. Participants with SCLC with prior treatment with stereotactic radiosurgery or whole brain radiation therapy for CNS metastatic disease 2 weeks or more before study start may be considered eligible for enrollment if assessed stable and meet all other eligibility criteria.
* History of stroke or intracranial hemorrhage within ≤6 months
* History of seizure or seizure disorder, ie, recurrent seizures with an underlying etiology and requiring ongoing anti-epileptic medication
* Current use of medications associated with seizure risk
* Active infections requiring systemic antibiotic, antiviral or antifungal therapy
* Known active coronavirus disease 2019 (COVID-19)
* Clinically significant heart disease
* Uncontrolled hypertension
* Prolongation of QT interval at baseline
* Known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Incidence of Adverse Events (AEs) | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 38 months)
  Type, incidence, severity, causality and outcome of adverse events (AEs), including serious AEs and AEs at Grade 3 or above, based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.
Part 1 and Part 2: Number of Participants with Dose Limiting Toxicity (DLT) of KB-0742 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days
Part 1: Maximally Tolerated Dose (MTD) of KB-0742 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days
Part 1: Recommended Phase 2 Dose (RP2D) of KB-0742 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days

SECONDARY OUTCOMES:
Part 1: Maximal Plasma Concentration (Cmax) of KB-0742 | Cycle 1 Day 1 through Cycle 6 Day 1, where a cycle is up to 28 days
Part 1: Time to Maximal Plasma Concentration (Tmax) of KB-0742 | Cycle 1 Day 1 through Cycle 6 Day 1, where a cycle is up to 28 days
Part 1: Area Under The Plasma Concentration x Time Curve From Hour 0 to The Last Measurable Time Point (AUC0-last) of KB-0742 | Cycle 1 Day 1 through Cycle 6 Day 1, where a cycle is up to 28 days
Part 1 and Part 2: Progression Free Survival (PFS) | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 38 months)
Part 1 and Part 2: Disease Control Rate | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 38 months)
Part 1 and Part 2: Duration of Disease Control | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 38 months)
Part 1 and Part 2: Overall Response Rate (ORR) | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 38 months)
Part 1 and Part 2: Duration of Response (DOR) | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 38 months)
Part 2: Maximal Plasma Concentration (Cmax) of KB-0742 | Cycle 1 Day 1 and Cycle 1 Day 12, where a cycle is up to 28 days
Part 2: Time to Maximal Plasma Concentration (Tmax) of KB-0742 | Cycle 1 Day 1 and Cycle 1 Day 12, where a cycle is up to 28 days
Part 2: Trough Concentration (Ctrough) of KB-0742 | Cycle 1 Day 1 and Cycle 1 Day 12, where a cycle is up to 28 days

CONTACTS AND LOCATIONS:
Locations (24):
- United States (20):
  - O'Neal Comprehensive Cancer Center at the University of Alabama, Birmingham, Alabama
  - City of Hope, Duarte, California
  - MemorialCare - Orange Coast Medical Center, Fountain Valley, California
  - City of Hope - Orange County Lennar Foundation Cancer Center, Irvine, California
  - Precision NextGen Oncology, Los Angeles, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Community Health Network Community Cancer Center South, Indianapolis, Indiana
  - Community Health Network Community Cancer Center North, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - Pennsylvania Cancer Specialists Research Institute - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - SCRI Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
- Sarah Cannon Research Institute London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No